CLINICAL TRIAL: NCT02433366
Title: Post-authorisation Study to Evaluate the Effectiveness of the Risk Minimisation Activities in the Treatment of SPAF
Brief Title: Evaluation the Effectiveness of the Risk Minimisation Activities in the Treatment of Stroke Prevention in Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.149
Record Dates: First submitted 2015-03-25; First posted 2015-05-05 (Estimated); Results first posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Patients
- Physicians

SUMMARY:
The key focus of this survey will be to collect data on physicians awareness of the content of the Pradaxa® Prescriber Guide and the extent to which risk awareness is communicated to patients. The data collected with atrial fibrillation patients will show if and how well this information is received and understood.

DETAILED DESCRIPTION:
Purpose:

ELIGIBILITY:
Inclusion criteria:

* Pradaxa® prescribers (cardiologists and primary care physicians)
* Patients with atrial fibrillation treated with Pradaxa®

Exclusion criteria:

As defined in Summary of Product Characteristics for patients treated with Pradaxa®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physicians prescribing dabigatran for patients with atrial fibrillation
Sampling Method: Probability Sample
Enrollment: 1213 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (161):
- Bulgaria (10):
  - Boehringer Ingelheim Investigational Site 81, Dobrich
  - Boehringer Ingelheim Investigational Site 84, Gabrovo
  - Boehringer Ingelheim Investigational Site 79, Montana
  - Boehringer Ingelheim Investigational Site 85, Plovdiv
  - Boehringer Ingelheim Investigational Site 80, Shumen
  - Boehringer Ingelheim Investigational Site 86, Sliven
  - Boehringer Ingelheim Investigational Site 87, Sofia
  - Boehringer Ingelheim Investigational Site 88, Stara Zagora
  - Boehringer Ingelheim Investigational Site 82, Varna
  - Boehringer Ingelheim Investigational Site 83, Veliko Tarnovo
- Czechia (29):
  - Boehringer Ingelheim Investigational Site 92, ?eská Lípa
  - Boehringer Ingelheim Investigational Site 93, ?eské Bud?jovice
  - Boehringer Ingelheim Investigational Site 94, ?eský Krumlov
  - Boehringer Ingelheim Investigational Site 90, B?eclav
  - Boehringer Ingelheim Investigational Site 89, Benesov U Prahy
  - Boehringer Ingelheim Investigational Site 91, Brno
  - Boehringer Ingelheim Investigational Site 95, Chomutov
  - Boehringer Ingelheim Investigational Site 96, Domažlice
  - Boehringer Ingelheim Investigational Site 97, Haví?ov
  - Boehringer Ingelheim Investigational Site 98, Havlí?k?v Brod
  - Boehringer Ingelheim Investigational Site 99, Ho?ovice
  - Boehringer Ingelheim Investigational Site 100, Hradec Králové
  - Boehringer Ingelheim Investigational Site 101, Ivan?ice
  - Boehringer Ingelheim Investigational Site 102, Krom??íz
  - Boehringer Ingelheim Investigational Site 103, Kyjov
  - Boehringer Ingelheim Investigational Site 104, Liberec
  - Boehringer Ingelheim Investigational Site 105, Louny
  - Boehringer Ingelheim Investigational Site 106, Most
  - Boehringer Ingelheim Investigational Site 107, Nový Bor
  - Boehringer Ingelheim Investigational Site 108, Odry
  - Boehringer Ingelheim Investigational Site 109, Olomouc
  - Boehringer Ingelheim Investigational Site 110, Pardubice
  - Boehringer Ingelheim Investigational Site 111, Plze?
  - Boehringer Ingelheim Investigational Site 112, Prague
  - Boehringer Ingelheim Investigational Site 113, Sternberk
  - Boehringer Ingelheim Investigational Site 114, Tábor
  - Boehringer Ingelheim Investigational Site 115, Tehovec
  - Boehringer Ingelheim Investigational Site 116, Teplice
  - Boehringer Ingelheim Investigational Site 117, Valasské Mezi?í?í
- Boehringer Ingelheim Investigational Site 69, Copenhagen, Denmark
- France (45):
  - Boehringer Ingelheim Investigational Site 25, Ambleuteuse
  - Boehringer Ingelheim Investigational Site 68, Ardres
  - Boehringer Ingelheim Investigational Site 26, Arnac-Pompadour
  - Boehringer Ingelheim Investigational Site 27, Audincourt
  - Boehringer Ingelheim Investigational Site 28, Bart
  - Boehringer Ingelheim Investigational Site 29, Besançon
  - Boehringer Ingelheim Investigational Site 30, Buissière Galant
  - Boehringer Ingelheim Investigational Site 31, Charbrignac
  - Boehringer Ingelheim Investigational Site 32, Châlus
  - Boehringer Ingelheim Investigational Site 33, Coussac-Bonneval
  - Boehringer Ingelheim Investigational Site 34, Décines-Charpieu
  - Boehringer Ingelheim Investigational Site 35, Eckwersheim
  - Boehringer Ingelheim Investigational Site 36, Geneuille
  - Boehringer Ingelheim Investigational Site 37, Glandon
  - Boehringer Ingelheim Investigational Site 65, Gruson
  - Boehringer Ingelheim Investigational Site 38, Halluin
  - Boehringer Ingelheim Investigational Site 39, Lanouaille
  - Boehringer Ingelheim Investigational Site 67, Le Catelet
  - Boehringer Ingelheim Investigational Site 40, Le Haillan
  - Boehringer Ingelheim Investigational Site 41, Lille
  - Boehringer Ingelheim Investigational Site 42, Limoges
  - Boehringer Ingelheim Investigational Site 43, Lomme
  - Boehringer Ingelheim Investigational Site 44, Lyon
  - Boehringer Ingelheim Investigational Site 45, Marseille
  - Boehringer Ingelheim Investigational Site 46, Mérignac
  - Boehringer Ingelheim Investigational Site 47, Nexon
  - Boehringer Ingelheim Investigational Site 48, Noaillan
  - Boehringer Ingelheim Investigational Site 24, Paris
  - Boehringer Ingelheim Investigational Site 52, Saint Saud Lacousserie
  - Boehringer Ingelheim Investigational Site 55, Saint-Hilaire-les-Places
  - Boehringer Ingelheim Investigational Site 50, Saint-Martial-d'Albarède
  - Boehringer Ingelheim Investigational Site 51, Saint-Martin-Sepert
  - Boehringer Ingelheim Investigational Site 53, Saint-Sornin-Lavolps
  - Boehringer Ingelheim Investigational Site 54, Saint-Yrieix-la-Perche
  - Boehringer Ingelheim Investigational Site 56, Schiltigheim
  - Boehringer Ingelheim Investigational Site 57, Sochaux
  - Boehringer Ingelheim Investigational Site 58, Strasbourg
  - Boehringer Ingelheim Investigational Site 59, Talence
  - Boehringer Ingelheim Investigational Site 60, Thiviers
  - Boehringer Ingelheim Investigational Site 66, Tourcoing
  - Boehringer Ingelheim Investigational Site 61, Tourmignies
  - Boehringer Ingelheim Investigational Site 49, Val Pompadour
  - Boehringer Ingelheim Investigational Site 62, Villenave-d'Ornon
  - Boehringer Ingelheim Investigational Site 63, Voujeaucourt
  - Boehringer Ingelheim Investigational Site 64, Weyersheim
- Germany (14):
  - Boehringer Ingelheim Investigational Site 9, Berlin
  - Boehringer Ingelheim Investigational Site 3, Bremen
  - Boehringer Ingelheim Investigational Site 10, Chemnitz
  - Boehringer Ingelheim Investigational Site 5, Düsseldorf
  - Boehringer Ingelheim Investigational Site 6, Essen
  - Boehringer Ingelheim Investigational Site 1, Frankfurt
  - Boehringer Ingelheim Investigational Site 8, Hanover
  - Boehringer Ingelheim Investigational Site 14, Heidelberg
  - Boehringer Ingelheim Investigational Site 11, Leipzig
  - Boehringer Ingelheim Investigational Site 2, Mannheim
  - Boehringer Ingelheim Investigational Site 7, Marburg
  - Boehringer Ingelheim Investigational Site 13, München
  - Boehringer Ingelheim Investigational Site 4, Nuremberg
  - Boehringer Ingelheim Investigational Site 12, Rostock
- Slovakia (44):
  - Boehringer Ingelheim Investigational Site 122, Banská Bystrica
  - Boehringer Ingelheim Investigational Site 127, Bardejov
  - Boehringer Ingelheim Investigational Site 152, Bratislava
  - Boehringer Ingelheim Investigational Site 146, Čierna nad Tisou
  - Boehringer Ingelheim Investigational Site 149, Čierne Kľačany
  - Boehringer Ingelheim Investigational Site 154, Čierny Brod
  - Boehringer Ingelheim Investigational Site 139, Dolné Kočkovce
  - Boehringer Ingelheim Investigational Site 141, Horný Vadičov
  - Boehringer Ingelheim Investigational Site 137, Ivanka pri Dunaji
  - Boehringer Ingelheim Investigational Site 140, Jelka
  - Boehringer Ingelheim Investigational Site 159, Kokava nad Rimavicou
  - Boehringer Ingelheim Investigational Site 125, Košice
  - Boehringer Ingelheim Investigational Site 158, Košťany nad Turcom
  - Boehringer Ingelheim Investigational Site 160, Krásno nad Kysucou
  - Boehringer Ingelheim Investigational Site 134, Lalinok
  - Boehringer Ingelheim Investigational Site 120, Lastovce
  - Boehringer Ingelheim Investigational Site 155, Liptovský Hrádok
  - Boehringer Ingelheim Investigational Site 145, Lučenec
  - Boehringer Ingelheim Investigational Site 144, Nitra
  - Boehringer Ingelheim Investigational Site 119, Nové Mesto nad Váhom
  - Boehringer Ingelheim Investigational Site 150, Nové Zámky
  - Boehringer Ingelheim Investigational Site 124, Odorín
  - Boehringer Ingelheim Investigational Site 142, Oščadnica
  - Boehringer Ingelheim Investigational Site 157, Poprad
  - Boehringer Ingelheim Investigational Site 128, Považská Bystrica
  - Boehringer Ingelheim Investigational Site 132, Považský Chlmec
  - Boehringer Ingelheim Investigational Site 118, Prešov
  - Boehringer Ingelheim Investigational Site 138, Púchov
  - Boehringer Ingelheim Investigational Site 143, Radoľa
  - Boehringer Ingelheim Investigational Site 153, Rešov
  - Boehringer Ingelheim Investigational Site 156, Revúca
  - Boehringer Ingelheim Investigational Site 147, Rožkovany
  - Boehringer Ingelheim Investigational Site 131, Rudinka
  - Boehringer Ingelheim Investigational Site 126, Sabinov
  - Boehringer Ingelheim Investigational Site 161, Skalité
  - Boehringer Ingelheim Investigational Site 123, Spišská Nová Ves
  - Boehringer Ingelheim Investigational Site 130, Stráňavy
  - Boehringer Ingelheim Investigational Site 121, Trebišov
  - Boehringer Ingelheim Investigational Site 151, Trnava
  - Boehringer Ingelheim Investigational Site 129, Trnové
  - Boehringer Ingelheim Investigational Site 135, Valasska Bela
  - Boehringer Ingelheim Investigational Site 148, Vráble
  - Boehringer Ingelheim Investigational Site 136, Zvolen
  - Boehringer Ingelheim Investigational Site 133, Žilina
- Spain (9):
  - Boehringer Ingelheim Investigational Site 23, Baleares
  - Boehringer Ingelheim Investigational Site 22, Barcelona
  - Boehringer Ingelheim Investigational Site 15, Ciudad Real
  - Boehringer Ingelheim Investigational Site 16, Galicia
  - Boehringer Ingelheim Investigational Site 17, Madrid
  - Boehringer Ingelheim Investigational Site 18, Murcia
  - Boehringer Ingelheim Investigational Site 19, Seville
  - Boehringer Ingelheim Investigational Site 20, Valencia
  - Boehringer Ingelheim Investigational Site 21, Zaragoza
- United Kingdom (9):
  - Boehringer Ingelheim Investigational Site 71, Brighton
  - Boehringer Ingelheim Investigational Site 76, Cheadle
  - Boehringer Ingelheim Investigational Site 78, Essex
  - Boehringer Ingelheim Investigational Site 70, London
  - Boehringer Ingelheim Investigational Site 77, Manchester
  - Boehringer Ingelheim Investigational Site 74, Middlesex
  - Boehringer Ingelheim Investigational Site 73, Romford
  - Boehringer Ingelheim Investigational Site 75, Stockport
  - Boehringer Ingelheim Investigational Site 72, Surrey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a cross-sectional survey. Pradaxa® prescribing healthcare professionals and Pradaxa® treated patients were randomly selected and interviewed (face-to-face).
  411 healthcare professionals and 802 patients with atrial fibrillation were enrolled and entered the study
Groups:
- Physicians: Current prescribers of Pradaxa® for stroke prevention in patients with atrial fibrillation (AF).
- Patients: AF patients on treatment with Pradaxa®.
Period: Overall Study
Arm/Group | Physicians | Patients
Started | 411 | 802
Completed | 411 | 802
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Physicians who were current prescribers of Pradaxa® for stroke prevention in patients with atrial fibrillation (AF) and AF patients who were currently receiving treatment with Pradaxa® entered this non-interventional survey
Groups:
- Total: Total of all reporting groups
Arm/Group | Physicians | Patients | Total
Number analyzed (Participants) | 411 | 802 | 1213
Age, Customized [Number; unit: Participants]
  <75 years | NA — Information about physicians age is not available | 480 | NA — Total not calculated because data are not available (NA) in one or more arms.
  ≥ 75 years | NA — Information about physicians age is not available | 322 | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Information about physicians gender is not available | 370 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Information about physicians gender is not available | 432 | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Physician's Knowledge and Recommendations to Their Patients on Appropriate Dosing and Minimizing the Risk of Bleeding When Treated With Pradaxa® (Questionnaire)
Description: The Outcome measure is summarized using the following categories; A: Physicians who spontaneously remembered the receipt of the Patient alert card, B: Physicians who spontaneously remembered the receipt of the Prescriber Guide, C: Physicians who were satisfied with the information provided in the Prescriber guide, D: Physicians who were aware of the importance of determining and controlling of the Patients renal function for correct pradaxa dosing.
  This Outcome measure is applicable only for the Physicians group.
Time Frame: Day 1
Population: Physicians who were current prescribers of Pradaxa® for stroke prevention in patients with atrial fibrillation (AF)
Measure: Number; unit: Percentage of Participants
Arm/Group | Physicians | Patients
Number analyzed (Participants) | 411 | 0
Percentage of Participants
  A | 65 |
  B | 71 |
  C | 95 |
  D | 100 |

2. Primary Outcome: Patient's Understanding of the Disease, Bleeding Signs, What to do in Case of Bleeding and How to Deal With Emergency Situations (Measuring Physician Compliance From Patient Perspective) (Questionnaire)
Description: The Outcome measure is summarized using the following categories; A: Patients who received the Patient Alert Card, read it and understood its content, B: Patients who completed the Patient Alert Card with the patient specific information, C: Patients who were well informed about their treatment and the actions to be taken in case of serious complications, D: Patents who knew about the anticoagulant effect of Pradaxa®, E: Patients who were well aware of the potential side effect-bruising, F: Patients who were well aware of the potential side effect-bleeding. This Outcome measure is applicable only for the Patients group.
Time Frame: Day 1
Population: AF patients on treatment with Pradaxa®.
Measure: Number; unit: Percentage of Participants
Arm/Group | Physicians | Patients
Number analyzed (Participants) | 0 | 802
Percentage of Participants
  A |  | 55
  B |  | 83
  C |  | 100
  D |  | 89
  E |  | 54
  F |  | 52

ADVERSE EVENTS:
Description: Adverse events (AE) were not reported in this trial report but in case a physician or patient mentioned an AE during the interview, the interviewer together with the physician or patient was to complete an AE form which was forwarded to pharmacovigilance unit of BI.
Arm/Group | Physicians | Patients
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights